CLINICAL TRIAL: NCT06569095
Title: Predictive Value of Myelodysplastic Syndrome Stem Cells Determined by Multiparameter Flow Cytometry in Patients Receiving Allotransplantation: a Multi-center, Prospective Clinical Study
Brief Title: Predictive Value of Myelodysplastic Syndrome Stem Cells Determined by Multiparameter Flow Cytometry
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Chinese PLA General Hospital (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Principal Investigator, Chang Yingjun, Professor and Chief Physician, Peking University People's Hospital
Other Study IDs: PekingUPH Chang YJ
Record Dates: First submitted 2024-07-15; First posted 2024-08-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MDS-EB
  Interventions: Other: Detection of MDS-SC using MFC

INTERVENTIONS:
Other: Detection of MDS-SC using MFC — The aim of this study is to investigate the predictive values of MDS-SC determined by MFC for patients with MDS-EB who underwent allotransplantation.

SUMMARY:
Presently, multiparameter flow cytometry (MFC) and polymerase chain reaction (PCR) have been used for disease load, including measurable residual disease (MRD), monitoring in patients with myelodysplastic syndrome (MDS). MFC is the most commonly method for disease load evaluation. In patients with acute myeloid leukemia, leukemia stem cells (LSCs) determined using MFC for leukemia load and MRD detection is superior to traditional MFC method. In the investigators previous single center study, the investigators demonstrated that detection of disease load, including MRD, by MFC in patients with MDS-EB is superior to predict outcomes after allogeneic stem cell transplantation. Here, the investigators will perform a multi-center, prospective clinical trial to investigate the predictive values of MDS-SC in patients with MDS-EB who received allografting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Myelodysplastic syndromes;
* Between 15 and 70 years old;
* Subjects are able to provide written informed consent.

Exclusion Criteria:

* Subjects who cannot comply with the study;
* Patient has severe cardiac (ejection fraction <50%), hepatic (total bilirubin >34μmol/L, ALT, AST >2x upper limit of normal) or renal (blood creatinine >130μmol/L) disease；
* Uncontrolled serious infection;
* Other conditions that do not tolerate transplantation or other therapies.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To determine whether there was any difference in relapse between the pre-transplant MRD-positive and -negative groups, the cumulative incidence approach was used with a test for equivalence of CIF for the difference in the Kaplan-Meier estimate of the 1-year CIR. With a planned sample size of 163 AML/MDS patients, 80% power can be achieved against the hypothesis of CIR as 18.3% and 3.6% for cases in the pre-transplant MRD-positive and -negative groups at a significance level of P = 0.05 in Student's one-tailed t-test.
Sampling Method: Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
1 year-cumulative relapse rate | through study completion, an average of 1 year
  Relapse was defined by the morphological evidence of disease in the peripheral blood, BM or extramedullary sites. Time to relapse was defined from the date of transplantation to the date of disease recurrence. Patients exhibiting minimal residual disease were not classified as having relapsed.

SECONDARY OUTCOMES:
Cumulative positive rate of measurable residual disease (MRD) after transplantation | through study completion, an average of 1 year
  The proportion of MRD positive patients after treatment.
Disease-free survival (LFS) | through study completion, an average of 1 year
  Disease-free survival was defined as days from transplantation to disease progression after transplantation.
Overall survival (OS) | through study completion, an average of 1 year
  Overall survival referred to patients who survived until the final follow-up time point.
Non-recurrent death (NRM) | through study completion, an average of 1 year
  Non-recurrent mortality was defined as all causes of death other than those related directly to malignant disease itself, occurring at any time after CR.
Transplant-related death (TRM) | through study completion, an average of 1 year
  Transplant-related death was defined as all causes of death other than those related directly to malignant disease itself, occurring at any time after transplantation.
Acute graft-versus-host disease (GVHD) | through study completion, an average of 1 year
  Acute GVHD was defined and graded from 0 to IV based on the pattern and severity of organ involvement; grades III-IV aGVHD manifest as serious clinical features on the skin, liver and/or gut.
Chronic graft-versus-host disease (GVHD) | through study completion, an average of 1 year
  Chronic GVHD was defined and graded according to the National Institute of Health criteria:[Biol Blood Marrow Transplant,2005,11: 945] that is, mild cGVHD reflects the involvement of no more than 1 or 2 organs/sites (except for lung) with a maximum score of 1; moderate cGVHD involves at least 1 organ/site with a score of 2 or ≥3 organs/sites with a score of 1 (or lung score 1); and severe cGVHD is diagnosed when a score of 3 is given to any organ (or lung score 2). The diagnosis is mainly based on clinical manifestations.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chinese PLA General Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Wuhan TongJi Hospital, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No